CLINICAL TRIAL: NCT04420650
Title: Improving Insulin Sensitivity by Non-invasive Brain Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: German Center for Diabetes Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: BRAINSTIM
Record Dates: First submitted 2020-05-26; First posted 2020-06-09 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-09

CONDITIONS: Insulin Resistance; Transcranial Direct Current Stimulation; Obesity; Diabetes; Magnetic Resonance Imaging
MeSH Terms: conditions — Insulin Resistance; Obesity; Diabetes Mellitus | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Anodal tDCS (Active Comparator): Anodal tDCS of the hypothalamus-cognitive network
  Interventions: Device: transcranial direct current stimulation
- Cathodal tDCS (Active Comparator): Cathodal tDCS of the hypothalamus-cognitive network
  Interventions: Device: transcranial direct current stimulation
- Sham Stimulation (Sham Comparator): Double blind sham stimulation (ramp-up ramp-down stimulation will be applied in order to simulate the active condition without any further continuous administration of current)
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — anodal or cathodal transcranial direct current stimulation

SUMMARY:
Efforts in curing and preventing obesity and type 2 diabetes (T2D) have been elusive thus far. One reason for that is the lack of understanding of the role of the brain in the development and treatment of the disease. In recent studies, the hypothalamus was identified as part of a brain network including higher cognitive regions that is particularly vulnerable to insulin resistance. Furthermore, the central insulin response in this network predicted food craving and hunger. In this project, transcranial direct current stimulation (tDCS) is implemented as a tool to stimulate brain networks. The investigators hypothesize that stimulating the hypothalamus-cognitive network will enhance insulin sensitivity and reduce food intake, food craving and hunger. Furthermore, the project will provide the unique opportunity to investigate novel mechanisms of insulin resistance in participants who have been extensively metabolically characterized.

DETAILED DESCRIPTION:
Objectives The overarching aim of the study is to stimulate the hypothalamus-cognitive brain network to improve insulin sensitivity and eating behavior.

Specific Objectives

1. Implement tDCS stimulation compared to sham stimulation in overweight and obese adults to assess the impact on eating behavior, cognition and metabolism.
2. Evaluate whether 3-day non-invasive brain stimulation of the hypothalamus-cognitive network has a causal effect on metabolism.
3. Evaluate whether 3-day non-invasive brain stimulation has a significant effect on brain functional connectivity and diffusion parameters.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 25.5 and 39.5 kg/m2
* Age between 20 to 66 years of age
* Waist circumference ≥ 80 cm for women, ≥ 94 cm for men

Exclusion Criteria:

* Insufficient knowledge of the German language
* Persons who cannot legally give consent
* Pregnancy or lactation
* History of severe mental or somatic disorders including neurological diseases (incl. epileptic seizures)
* Taking psychotropic drugs
* Previous bariatric surgery
* Acute infection within the last 4 weeks
* Hemoglobin values less than 12g/dl for women, less than 14 g/dl for men
* Current participation in a lifestyle intervention study or a pharmaceutical study
* Contradictions to a MRI measurement (e.g. metal implants)

Ages: 20 Years to 66 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-05-26 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-11-10 (Actual)

PRIMARY OUTCOMES:
Peripheral insulin sensitivity | 1 day after last intervention tDCS day
  Oral glucose tolerance derived insulin sensitivity based on the Matsuda index
Caloric intake (kcal) | 1 hour directly after tDCS stimulation
  Free-choice, ad libitum food intake from a standardized breakfast buffet. The caloric intake from fat, carbohydrates and protein will be documented.
Change in subjective feeling of hunger and food craving | 5 minutes before tDCS stimulation, 5 minutes after tDCS stimulation and 5 minutes after buffet
  On a visual analogue scale, subjective feeling of hunger and food craving will be assessed using a questionnaire.

SECONDARY OUTCOMES:
Performance during stop-signal task | task is performed during 25-minutes tDCS stimulation
  Outcome measures cover direction errors, proportion of successful stops, reaction time on Go trials, and stop signal reaction time (SSRT).
Tastiness and healthiness rating of food stimuli | task is performed immediatly after buffet
  Using a computer based task, participants rate food pictures of low caloric and high caloric foods and snacks on a 5-point scale based on subjective tastiness and healthiness.
Food choice | task is performed immediatly after buffet
  Using a computer based task, participants have to choose food items they preferred to eat compared to a reference food on a 5-point choice scale. The reference (or "neutral") food item is individually determined based the health and taste rating [Scale: 1= not tasty/ not healthy up to 5= very tasty/ very heahlty].
Functional connectivity | 10 minutes functional MRI measurement performed before and after three day tDCS stimulation
  Resting-state functional connectivity of the hypothalamus-cognitive network is assessed by functional magnetic resonance imaging (fMRI)
Diffusion-weighted imaging | 15 minutes MRI measurement performed before and after three day tDCS stimulation
  Diffusion weighted parameter based on MRI measurements

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Kullmann, PhD, Principal Investigator — Univeristy of Tübingen, Germany
Locations (1):
- University Clinic Tübingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No